CLINICAL TRIAL: NCT02563509
Title: Reconstitution of HIV-specific Immunity Against HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou 8th People's Hospital (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Linghua LI, Chief physician, Guangzhou 8th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013ZX10001004
Record Dates: First submitted 2015-09-13; First posted 2015-09-30 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: HIV
Keywords: HIV; cellular immunity therapy; functional cure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-specific CD8 cells (Experimental): Transfusing HIV-specific CD8 cells 50-100mlonce a week for four times.
  Interventions: Biological: HIV-specific CD8 cells
- Regualar therapy (No Intervention): Only receiving Highly active anti-retroviral therapy(HAART).

INTERVENTIONS:
Biological: HIV-specific CD8 cells — Based on HAART, receive HIV-specific CD8 cells transfuion.
  Arms: HIV-specific CD8 cells

SUMMARY:
Research Goal: To reconstitute the anti-HIV specific immunity system of the AIDS patients, so the viruses could not massively replicate when HAART was discontinued, then make HIV functional cure possible.

DETAILED DESCRIPTION:
The research aims at establishing a new treatment strategies of HIV. It will significantly improve the clinical therapy effects and effectively reduce the morbidity and mortality by reconstituting the immune systems of HIV infected patients and combining multiple therapy strategies. Therefore, the research could develop an cloning amplification system of immunocytes in vitro, and improve the antiviral immune system severely damaged before by transfusing the clone cells modified by specific HIV antigen. So HIV infected patients could discontinue the traditional anti-viral drug, but not develop opportunistic infections,which could obviously increase the life qualities of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection confirmed
2. Receiving HAART more than 6 months
3. HIV viral-load < 50 copies/ml
4. Without serious damage of liver and kidney
5. The subject volunteered to the research and sign the informed consent

Exclusion Criteria:

1. With serious opportunistic infections
2. With serious chronic disease such like diabetes, the mental illness,et al
3. History of suffering from pancreatitis during HAART.
4. Pregnant and breast-fed.
5. With poor adherence

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The number and function of HIV-specific CD8 cells in patients with HIV | 6 Months
  The change of differentiation, proliferation, apoptosis, phenotype, etal.

SECONDARY OUTCOMES:
All adverse events | 6 Months
  Chills, Fever, Headache, Nausea, Vomiting, Cough, Skin rashes, Anaphylactic shock, Etal.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhang, doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Guangzhou 8th People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fidler S, Olson A, Fox J, Phillips A, Morrison C, Thornhill J, Bucher H, Muga R, Porter K. The importance of viral blips and duration of therapy initiated in primary infection in maintaining viral control after stopping cART. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19820. doi: 10.7448/IAS.17.4.19820. eCollection 2014. PMID 25397564
- [Background] Archin NM, Sung JM, Garrido C, Soriano-Sarabia N, Margolis DM. Eradicating HIV-1 infection: seeking to clear a persistent pathogen. Nat Rev Microbiol. 2014 Nov;12(11):750-64. doi: 10.1038/nrmicro3352. PMID 25402363
- [Background] Chew N, Tan E, Li L, Lim R. HIV-1 tat and rev upregulates osteoclast bone resorption. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19724. doi: 10.7448/IAS.17.4.19724. eCollection 2014. PMID 25397470
- [Background] Abdel-Mohsen M, Deng X, Danesh A, Liegler T, Jacobs ES, Rauch A, Ledergerber B, Norris PJ, Gunthard HF, Wong JK, Pillai SK. Role of microRNA modulation in the interferon-alpha/ribavirin suppression of HIV-1 in vivo. PLoS One. 2014 Oct 2;9(10):e109220. doi: 10.1371/journal.pone.0109220. eCollection 2014. PMID 25275557
- [Background] Vandergeeten C, Fromentin R, DaFonseca S, Lawani MB, Sereti I, Lederman MM, Ramgopal M, Routy JP, Sekaly RP, Chomont N. Interleukin-7 promotes HIV persistence during antiretroviral therapy. Blood. 2013 May 23;121(21):4321-9. doi: 10.1182/blood-2012-11-465625. Epub 2013 Apr 15. PMID 23589672
- [Background] Cahn P, Ruxrungtham K, Gazzard B, Diaz RS, Gori A, Kotler DP, Vriesema A, Georgiou NA, Garssen J, Clerici M, Lange JM; (BTE) Blinded Nutritional Study for Immunity and Tolerance Evaluation Study Team. The immunomodulatory nutritional intervention NR100157 reduced CD4+ T-cell decline and immune activation: a 1-year multicenter randomized controlled double-blind trial in HIV-infected persons not receiving antiretroviral therapy (The BITE Study). Clin Infect Dis. 2013 Jul;57(1):139-46. doi: 10.1093/cid/cit171. Epub 2013 Mar 19. PMID 23511299
- [Result] Sandler NG, Bosinger SE, Estes JD, Zhu RT, Tharp GK, Boritz E, Levin D, Wijeyesinghe S, Makamdop KN, del Prete GQ, Hill BJ, Timmer JK, Reiss E, Yarden G, Darko S, Contijoch E, Todd JP, Silvestri G, Nason M, Norgren RB Jr, Keele BF, Rao S, Langer JA, Lifson JD, Schreiber G, Douek DC. Type I interferon responses in rhesus macaques prevent SIV infection and slow disease progression. Nature. 2014 Jul 31;511(7511):601-5. doi: 10.1038/nature13554. Epub 2014 Jul 9. PMID 25043006
- [Result] Bouchat S, Gatot JS, Kabeya K, Cardona C, Colin L, Herbein G, De Wit S, Clumeck N, Lambotte O, Rouzioux C, Rohr O, Van Lint C. Histone methyltransferase inhibitors induce HIV-1 recovery in resting CD4(+) T cells from HIV-1-infected HAART-treated patients. AIDS. 2012 Jul 31;26(12):1473-82. doi: 10.1097/QAD.0b013e32835535f5. PMID 22555163
- [Result] Crawford TQ, Hecht FM, Pilcher CD, Ndhlovu LC, Barbour JD. Activation associated ERK1/2 signaling impairments in CD8+ T cells co-localize with blunted polyclonal and HIV-1 specific effector functions in early untreated HIV-1 infection. PLoS One. 2013 Oct 15;8(10):e77412. doi: 10.1371/journal.pone.0077412. eCollection 2013. PMID 24143233